CLINICAL TRIAL: NCT02692274
Title: Evaluating the Accessibility and Utility of HIV-related Point of Care Diagnostic for Maternal Health in Rural South Africa
Brief Title: Operational Assessment of Point-of-Care Diagnostics in Primary Healthcare Clinics
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Collaborators: African Population and Health Research Center (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Tivani Mashamba-Thompson, Mrs, University of KwaZulu
Other Study IDs: BE484/14; HRKM 40/15 (Other: KwaZulu Natal Department of Health)
Record Dates: First submitted 2016-02-18; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: HIV
Keywords: Point-of-care diagnostics; Rural primary health care; Access; Need; Usage; Maternal Health

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for evaluating the accuracy of HIV rapid tests in rural KwaZulu Natal
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Health care clinics: A survey of 100 primary Health care clinics was carried out
- Pregnant and breast feeding women: 208 patients were recruited from nine clinics that participated in the survey for evaluation of the accuracy of results produced by the HIV rapid test.

SUMMARY:
Diagnostic point-of-care (POC) tests are being rapidly developed and implemented in resource-limited settings. There has been a rapid rise of HIV and TB POC tests in South Africa during the last 10-15 years. The investigators sought to determine the existing availability, current usage and future need of POC tests among rural primary healthcare (PHC) clinics in South Africa's KwaZulu-Natal Province.

DETAILED DESCRIPTION:
Several new diagnostics generation devices are specifically designed to assist clinical staff replacing the equivalent laboratory tests and allowing a wide range of disease diagnoses to be performed immediately at the POC. The clinical impact of POC diagnostics has been shown in a variety of diseases conditions, particularly HIV/AIDS and TB. The World Health Organisation (WHO) called for new clinical diagnostics methods that are designed to function in setting with limited access to laboratory services. Thus, leading to an increase in marketing, manufacturing and development of POC diagnostics instruments and reagents for use in clinical POC. The advent of POC tests in South Africa has led to an improved control of infectious diseases such as HIV and mycobacterium tuberculosis (TB), in this era of drug-resistance. Increased availability of POC test in rural and resource-limited settings is encouraged.

To maximize the impact of novel diagnostics on patient outcomes in resource-limited settings, the implementation of new diagnostics must be performed within a given context and culture. However, the population-level of diagnostic utility in South Africa is not known. The investigators aim to estimate the level of POC diagnostic availability, usage and need in rural South Africa, using a cross sectional survey of rural primary healthcare (PHC) clinics in KwaZulu Natal (KZN). The survey focused on the conditions for which the respondent considered a POC test might help improve their clinical decision making during patient care. Determining the current accessibility, availability, usage and need for POC diagnostics in rural and resource limited settings can help inform developers and implementers of POC diagnostic services on context-specific deployment and implementation of POC diagnostics to address the unmet needs of patients in these settings.

ELIGIBILITY:
Inclusion Criteria:

* Primary Healthcare clinics located in rural and semi-rural settings

Exclusion Criteria:

* Primary Healthcare clinics located in urban settings

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Rural Primary Healthcare clinics
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Accessibility and availability | Three months
  The accessibility and availability of point-of-care diagnostics for maternal health patients in rural primary healthcare clinics

SECONDARY OUTCOMES:
Usage | Three months
  The utility of point-of-care diagnostics for maternal health patients in rural South Africa

CONTACTS AND LOCATIONS:
Overall Officials: Tivani P Mashamba-Thompson, Masters, Principal Investigator — University of KwaZulu; Benn K Sartorius, PhD, Study Director — University of KwaZulu; Paul K Drain, MD,MPH, Study Director — University of Washington
Locations (1):
- University of KwaZulu Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drain PK, Garrett NJ. The arrival of a true point-of-care molecular assay-ready for global implementation? Lancet Glob Health. 2015 Nov;3(11):e663-4. doi: 10.1016/S2214-109X(15)00186-2. No abstract available. PMID 26475005
- [Background] Drain PK, Hyle EP, Noubary F, Freedberg KA, Wilson D, Bishai WR, Rodriguez W, Bassett IV. Diagnostic point-of-care tests in resource-limited settings. Lancet Infect Dis. 2014 Mar;14(3):239-49. doi: 10.1016/S1473-3099(13)70250-0. Epub 2013 Dec 10. PMID 24332389
- [Background] Nabyonga J, Orem J. From knowledge to policy: lessons from Africa. Sci Transl Med. 2014 Jun 11;6(240):240ed13. doi: 10.1126/scitranslmed.3008852. No abstract available. PMID 24920657
- [Background] Thomas TL, DiClemente R, Snell S. Overcoming the triad of rural health disparities: How local culture, lack of economic opportunity, and geographic location instigate health disparities. Health Educ J. 2014 May;73(3):285-294. doi: 10.1177/0017896912471049. PMID 25242822
- [Derived] Mashamba-Thompson TP, Sartorius B, Drain PK. Operational assessment of point-of-care diagnostics in rural primary healthcare clinics of KwaZulu-Natal, South Africa: a cross-sectional survey. BMC Health Serv Res. 2018 May 29;18(1):380. doi: 10.1186/s12913-018-3207-6. PMID 29843711